CLINICAL TRIAL: NCT03119935
Title: Evaluation of an Amflow-device Assist Ambu-bagging to Improve Accuracy of Tidal Volumes Delivered.
Brief Title: Amflow-device Can Help Proper Ambu-bag Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Amflow
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Ventilation Therapy; Complications
Keywords: ambu bag, ventilation, tidal volume
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amflow assist ambu bag ventiation (Experimental): Newely developed method (Amflow assist ambu bag ventilation)
  Interventions: Device: Amflow
- Ambu bag ventilation (Experimental): Ordinary method (ambu bag ventilation
  Interventions: Device: Ambu bag

INTERVENTIONS:
Device: Amflow — Amflow deviced was developed for monitoring ventiation rate and ventilation volume. Participants ventilated the simulated patients by Amflow-device assist ambu bag
  Arms: Amflow assist ambu bag ventiation
Device: Ambu bag — Participants ventilated the simulated patients by ambu bag
  Arms: Ambu bag ventilation

SUMMARY:
This is a simulation study with a prospective randomized cross-over design. The aim of this study is to evaluate whether Amflow-assisted ambu-bag can delivery the accurate tidal volume compare to ordinary ambu-bag

DETAILED DESCRIPTION:
Ambu-bag ventilation is an essential skill to the patients who needed ventilatory support. However, the delivery of appropriate amount of tidal volume by ordinary manual bag ventilation may be difficult. In addition, it require adequate training to rescurer.

We hypothesised that an Amflow assist ambu bag may be helpful to delivery accurate tidal volumes to the patients.

Participants performed bag-valve ventilation to manikin by ordinary technique and Amflow assist technique in our simulation centre. We measured each ventilation rate and ventilation volume in simulated scenario and we compare those between two technique.

ELIGIBILITY:
Inclusion Criteria:

* A healthy senior medical students who agree attend this study.

Exclusion Criteria:

* A participants who does not agree attend this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Tidal volume | 6 minutes
  We compared mean tidal volume delivered to manikins between two techniques

SECONDARY OUTCOMES:
Ventilation Rate | 6 minutes
  We compared mean ventilation rate between two techniques

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, Dr, Principal Investigator — Department of Emergency Medicine, School of Medicine, Konkuk University, Konkuk University Medical Center
Locations (1):
- Department of Emergency Medicine, Konkuk University Medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No